CLINICAL TRIAL: NCT01113203
Title: Chronic and Acute Effects of Resistance Exercise on Older Subjects' Blood Pressure
Acronym: RTBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Associacao Fundo de Incentivo a Psicofarmcologia (Other); Federal University of São Paulo (Other); Delboni Auriemo (Unknown)
Responsible Party: Cláudia Lúcia de Moraes Forjaz, School of Physical Education, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNPq471600/2008-3
Record Dates: First submitted 2010-04-27; First posted 2010-04-29 (Estimated); Last update posted 2010-04-29 (Estimated); Status verified 2010-04

CONDITIONS: Blood Pressure
Keywords: resistance training; blood pressure; hemodynamics; autonomic; Elderly Subjects
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Resistance training (Experimental): Progressive high intensity resistance training performed twice a week for 16 weeks, and achieving in 7 exercises for the main muscles, the protocol of 4 sets of 6RM and 2 of 4RM.
  Interventions: Behavioral: Resistance training

INTERVENTIONS:
Behavioral: Resistance training — Progressive high intensity resistance training performed twice a week for 16 weeks, and achieving in 7 exercises for the main muscles, the protocol of 4 sets of 6RM and 2 of 4RM.
  Other Names: strength training, weight training

SUMMARY:
The study aimed to evaluate the chronic and acute effects of high-intensity resistance training on blood pressure and its hemodynamic and neural determinators in healthy normotensive older subjects.

DETAILED DESCRIPTION:
To investigate the chronic and acute effects of resistance training on blood pressure and its hemodynamic and neural determinators in elderly, 24 healthy normotensive older subjects were randomly divided into 2 groups: trained and control. The trained group was submitted a progressive high-intensity resistance training. Before and after 16 weeks, as well as, before and after the one training session, blood pressure (clinic and ambulatory), cardiac output (CO2 rebreathing), and autonomic modulation (spectral analysis of heart rate and blood pressure variabilities) were measured

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 80 years
* Normotensives
* Nonactive

Exclusion Criteria:

* Cardiovascular disease
* Cardiovascular medication
* Orthopedic problems

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
blood pressure | 16 weeks
  Blood pressure was measured by auscultatory, oscillometric and photoplethysmographic device

SECONDARY OUTCOMES:
cardiovascular hemodynamics | 16 weeks
  cardiac output (CO2 rebreathing technique)
cardiovascular autonomic modulation | 16 weeks
  Spectral analysis of heart rate and blood pressure variabillity

CONTACTS AND LOCATIONS:
Overall Officials: Claudia LM Forjaz, PhD, Principal Investigator — School of Physical Education and Sport, University of São Paulo
Locations (1):
- School of Physical Education and Sport, University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Queiroz AC, Kanegusuku H, Chehuen MR, Costa LA, Wallerstein LF, Dias da Silva VJ, Mello MT, Ugrinowitsch C, Forjaz CL. Cardiac work remains high after strength exercise in elderly. Int J Sports Med. 2013 May;34(5):391-7. doi: 10.1055/s-0032-1323779. Epub 2012 Nov 22. PMID 23175179